CLINICAL TRIAL: NCT00225862
Title: A 12-week, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of Intermittent Dosing of Ropinirole in Patients With Restless Legs Syndrome (RLS)
Brief Title: A Clinical Research Study Evaluating Ropinirole Treatment For Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100310
Record Dates: First submitted 2005-06-30; First posted 2005-09-26 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Restless Legs Syndrome
Keywords: RLS; Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ropinirole

SUMMARY:
A 12-week clinical research study to evaluate the tolerability, efficacy and safety of ropinirole compared to placebo(an inactive sugar pill) in the treatment of patients with RLS in the United States.

ELIGIBILITY:
Â Inclusion criteria:

* Patients diagnosed with Restless Legs Syndrome (RLS).
* Patients diagnosed with RLS (symptoms include an overwhelming urge to move legs usually accompanied by uncomfortable sensations in the legs; usually occur at rest; worse during the evening or night and generally relieved, at least temporarily, by movement).
* Patients must give written informed consent prior to any specific study procedures.

Exclusion criteria:

* Patients with a primary sleep disorder other than RLS.
* Patients with symptoms of secondary RLS (i.e., renal failure, iron deficient anemia, pregnancy) or other movement disorders (i.e., Parkinson's Disease).
* Other inclusion or exclusion criteria to be evaluated by the physician.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-01; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Average proportion of nights a subject has successfully treated his/her RLS symptoms after taking study medication for that night out of total number of nights dosed during the Double-Blind Phase. | 12 Weeks

SECONDARY OUTCOMES:
Quality and satisfaction with sleep, severity of symptoms 2 hours post dosing with study medication. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (36):
- United States (36):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Fairfield, Connecticut
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Elk Grove Village, Illinois
  - GSK Investigational Site, Flossmoor, Illinois
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Frederick, Maryland
  - GSK Investigational Site, Newton, Massachusetts
  - GSK Investigational Site, Newton Center, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Amherst, New York
  - GSK Investigational Site, New Hyde Park, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Concinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Lafayette Hill, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Walla Walla, Washington
  - GSK Investigational Site, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 100310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 100310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100310 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register